CLINICAL TRIAL: NCT03793023
Title: Observational Study to Evaluate the Efficacy and Safety of Teneligliptin When Switched From Other DPP-4 Inhibitors in Type 2 DM With Inadequate Glycemic Control
Brief Title: Observational Study to Evaluate the Efficacy and Safety of Teneligliptin
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD_TEN_OS2015
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Teneligliptin 20mg

SUMMARY:
This study is designed as a prospective, observational, multi-centre study to evaluate the efficacy and safety of Teneligliptin when switched from other DPP-4 inhibitors in type 2 DM with inadequate glycemic control

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged ≥19 years
2. The subject has a documented diagnosis of type 2 diabetes mellitus for at least 3 months at the screening visit.
3. Patient who was treated with same dosage of DPP4 inhibitor for at least 12 weeks prior to baseline visit (if patient who has been treated with DPP4 inhibitor and any other antidiabetic drugs, antidiabetic drugs should also have been kept same dosage for at least 12 weeks prior to baseline.)
4. Patient with HbA1c≥7.0% at baseline visit
5. Patient who can be switched to Teneligliptin instead of using DPP-4 inhibitor for glycemic control based on the investigator's judgment
6. Patient (or legal guardian, if applicable) is informed of the full nature and purpose of the study, including possible risks and side effects, and understand this information, voluntarily signed and dated the written informed consent in compliance with protocol before inclusion in the study

Exclusion Criteria:

1. Patient with hypersensitivity to the Teneligliptin
2. Patient who treat the Teneligliptin prior to baseline visit
3. A pregnant or lactating female patient

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 2 DM patients
Sampling Method: Probability Sample
Enrollment: 2983 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | at 12 weeks after switching to Teneligliptin
  To assess change from baseline in glycated hemoglobin (HbA1c)

SECONDARY OUTCOMES:
Change in HbA1c | at 24, 52 weeks after switching to Teneligliptin
  To assess change from baseline in HbA1c
Change in FBG | at 12, 24, 52 weeks after switching to Teneligliptin
  To assess change from baseline in fasting blood glucose (FBG)
Change in body weight, BMI | at 12, 24, 52 weeks after switching to Teneligliptin
  To assess change from baseline in body weight and body mass index (BMI)
Change in lipid profile(Total cholesterol, LDL cholesterol, HDL cholesterol) | at 12, 24, 52 weeks after switching to Teneligliptin
  To assess change from baseline in serum lipid profile (total cholesterol, LDL and HDL cholesterol, triglyceride)
The percentage of patients with HbA1c <7.0% and <6.5% | at Weeks 12, 24, and 52 of teneligliptin treatment
  To assess the percentage of patients with HbA1c <7.0% and <6.5%
The percentage of patients with a decrease from baseline in HbA1c | at Weeks 12, 24, and 52 of teneligliptin treatment
  To assess the percentage of patients with a decrease from baseline in HbA1c by ≥0.3% and ≥ 0.5%
Safety Outcome | at Weeks 12, 24, and 52 of teneligliptin treatment
  To assess the safety of teneligliptin treatment(AE, ADR, SAE etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Kwan Woo Lee, MD, Ph.D, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Kim YS, Lee CB, Choi MG, Chang HJ, Kim SK, Yu JM, Kim TH, Lee JH, Ahn KJ, Kim K, Lee KW. Efficacy and Safety of Switching to Teneligliptin in Patients with Type 2 Diabetes Inadequately Controlled with Dipeptidyl Peptidase-4 Inhibitors: A 12-Week Interim Report. Diabetes Ther. 2019 Aug;10(4):1271-1282. doi: 10.1007/s13300-019-0628-0. Epub 2019 May 11. PMID 31079357